CLINICAL TRIAL: NCT03466034
Title: The Role of Hypoxia as a Selective Pressure for TP53 Mutations
Status: Terminated | Type: Observational
Why Stopped: Low numbers of eligible patients and failure to successfully recruit them.
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Principal Investigator, Nandita deSouza, Professor, Institute of Cancer Research, United Kingdom
Other Study IDs: CCR 4784
Record Dates: First submitted 2018-02-12; First posted 2018-03-15 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Endometrial Cancer
Keywords: TP53; Hypoxia; Endometriod and Mucinous Carcinomas; Serous and Clear Cell Carcinomas; Magnetic Resonance Imaging, MRI
MeSH Terms: conditions — Endometrial Neoplasms; Hypoxia; Adenocarcinoma, Mucinous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Endometrial tumour tissue Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endometriod: Type I (endometrioid and mucinous carcinomas) - Magnetic Resonance Imaging (MRI) with 100% Oxygen.
- Serous: Type II (serous and clear cell carcinomas) - Magnetic Resonance Imaging (MRI) with 100% Oxygen.

SUMMARY:
The study aims to develop scans that tell the investigators about the oxygen content of tumours using Magnetic Resonance Imaging (MRI) and seeing whether regions of low oxygen content are related to mutations in cancer genes such as TP53. MRI is a method of obtaining pictures of inside of the body that shows the appearance and structure of soft tissues.

To get the information about the oxygen content of tumours, MRI is carried out while breathing 100% oxygen. The variation of oxygen supply to different regions of the tumour will help the investigators to predict tumour behavior and tumour response to treatment.

DETAILED DESCRIPTION:
Cancer tissue harbours a multitude of genetic alterations, and it is well-established that when certain key alterations develop, they are powerful determinants of tumour behaviour (growth rate, potential to spread). One of the most sinister and well-recognized alterations is in a gene called TP53. Another feature of tumours that results in resistance to treatment and poor outcome is a low oxygen level within tumour tissue. However, whether alterations in TP53 are driven by low oxygen levels is not established.

Endometrial cancer is a good model to study the relationship between low tumour oxygen levels and alterations in TP53 within tumour. Firstly, it is a common gynaecological malignancy, (9,300 new cases annually in the UK) with two recognized types based on the appearance and behaviour of the tumour. In type I (endometrioid and mucinous carcinomas), alterations in TP53 are uncommon (15%), while in type II (serous and clear cell carcinomas) they are common (88%). In-line with this, the survival of patients with Type 2 cancer is worse. Secondly, endometrial cancer is routinely assessed at diagnosis using Magnetic Resonance Imaging. This non-invasive scanning technique can be manipulated to derive additional information about the oxygen status of the whole tumour and regions within it. Finally, the primary management of endometrial cancer is surgical and involves hysterectomy. This means it is possible to obtain fresh tumour tissue at the time of surgery from regions that have been identified on imaging as having low vs.high levels of oxygen and to establish their TP53 status. In this study, therefore, the investigator will establish the regional oxygen distribution within endometrial cancers at diagnosis, and relate them to the alterations in TP53 from fresh tissue samples from selected regions using gene sequencing. Understanding how highly deleterious mutations arise in cancer might provide new avenues for intervention and control.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age on the day of signing the informed consent.
2. Histologically confirmed endometroid or serous endometrial cancer.
3. Scheduled to have hysterectomy at the cancer centre
4. Identifiable tumour mass on staging MRI.
5. Voluntarily agreed to participate by giving written informed consent.

Exclusion Criteria:

1. Life expectancy of < 6 months.
2. Ferromagnetic implants, contraindicating MRI
3. Claustrophobia so unable to tolerate MRI
4. Unable to lie flat
5. Ascites sufficient to prevent patient being fitted in the scanner bore
6. Histology unlikely to show variation in TP53 status, or heavily calcified disease.
7. Radiotherapy to the abdomen or pelvis within 6 months of the screening visit.
8. Unresolved bowel obstruction.
9. Currently participating or has participated in a study with an investigational compound or device within 30 days of the start of treatment.
10. History or current evidence of any condition, therapy, or lab abnormality that might confound the results of the study, interfere with patient's participation for the full duration of the study, or is not in the best interest of the patient to participate.
11. Unlikely to comply with the requirements of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants scheduled to have hysterectomy at the cancer centre
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2018-06-19 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Establish distinctive patterns of distribution and expression of mutant TP53 between tumour regions with differing levels of oxygenation (as measured by R2*on MRI). | Duration of study (24 months)
  Determined at post surgery histology

SECONDARY OUTCOMES:
The reproducibility of the R2* measurement, assessed by comparing 2 R2* scans per person | 6 months
  comparison of image data at conclusion of MRI scan
Establish the range of intratumoral heterogeneity of the R2* measurement within individual tumours | 6 months
  comparison of image data at conclusion of MRI scan

CONTACTS AND LOCATIONS:
Overall Officials: Nandita deSouza, Principal Investigator — The Institution of Cancer Research & The Royal Marsden NHS Foundation Trust
Locations (1):
- The Institute of Cancer Research & The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom